CLINICAL TRIAL: NCT03536377
Title: Implementation of a Very Low Calorie Diet for Remission of Type 2 Diabetes in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDRS2
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Diabetes Mellitus Remission; Prediabetic State; caloric restriction; weight loss; diet; Barbados
MeSH Terms: conditions — Prediabetic State; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- very low calorie liquid diet (Experimental): Phase 1: Caloric restriction Phase 2: Solid diet Phase 3: Transition to independence
  Interventions: Other: very low calorie liquid diet

INTERVENTIONS:
Other: very low calorie liquid diet — Phase 1: very low calorie liquid formulation Phase 2: Nutritionally balanced solid diet Phase 3: Educational material

SUMMARY:
The complications associated with uncontrolled type-2 diabetes mellitus (T2DM) are numerous; reducing the quality of life for the patient and consuming a considerable portion of healthcare finances.

The Health of the Nation (HotN) 2011 study reported that 50% of the Barbadian population >65years old had a diagnosis of T2DM and that two-thirds of the population were overweight - which is a risk factor for the development of T2DM.

Encouraged by the success of the Counterpoint study in the United Kingdom (UK), the Barbados Diabetes Reversal Study 1 (BDRS1) was established using a similar protocol; the aim of which was to evaluate the feasibility of implementing a very low calorie diet to reverse T2DM in Barbados. At the end of the 8-week intervention period, the 25 participants had achieved an average weight loss of 10.1kg (22lbs). This was accompanied by an increase in the number of participants whose fasting blood sugars were now within normal range despite being off of their diabetes medication; and a decrease in the number of participants taking blood pressure medication. Participants transitioned to a solid diet over a 4-week period, with guidance on health dietary habits and regular exercise routines. The benefits accrued during the intervention phase were preserved at the end of the transition period.

We now propose the Barbados Diabetes Remission Study 2 (BDRS2) as a sustainable community intervention - utilizing the local church as the community site. We hypothesize that this will enhance reach while reducing the cost of the study and will also facilitate the structures necessary for the social support of the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 - 70 years old, all ethnicities
* Diagnosis of T2DM for <6 years as defined by the American Diabetes Association
* Diagnosis of pre-diabetes as defined by the American Diabetes Association
* Body Mass index (BMI) of 27 kg/m2 and over

Exclusion Criteria:

* Insulin use
* Substance abuse
* Current cancer diagnosis
* myocardial infarction within last 6 month
* learning difficulties
* current treatment with anti-obesity drugs
* diagnosed eating disorder or purging
* HbA1c > 10%
* pregnant/considering pregnancy
* evidence of liver disease (including liver enzymes > 3 times above normal values)
* evidence of renal disease (creatinine of > 150 mmol/l)
* persons who have required hospitalisation for depression, or are on antipsychotic drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change in weight | enrolment, 12 weeks, 6 mths and 1 year
change in fasting glucose | Enrolment, 12 weeks, 6 months, 1 year
change in Hba1C | Enrolment, 12 weeks, 6 months, 1 year

SECONDARY OUTCOMES:
change in waist circumference | Enrolment, 12 weeks, 6 months, 1 year
change in blood pressure | Enrolment, 12 weeks, 6 months, 1 year
  both the systolic and diastolic pressures will be measured
change in blood pressure medication | weekly for the first 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: T Alafia Samuels, MBBS, PhD, Study Chair — George Alleyne Chronic Disease Research Centre, The University of the West Indies
Locations (4):
- Barbados (4):
  - Abundant Life Assembly, Bridgetown, Bank Hall, Saint Michael
  - Ellerton Wesleyan Church, Bridgetown, Ellerton, Saint George
  - River Road New Testament Church of God, Bridgetown, River Road, Saint Michael
  - Mount of Praise Wesleyan Church, Bridgetown, Tudor Bridge, Saint Michael

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lim EL, Hollingsworth KG, Aribisala BS, Chen MJ, Mathers JC, Taylor R. Reversal of type 2 diabetes: normalisation of beta cell function in association with decreased pancreas and liver triacylglycerol. Diabetologia. 2011 Oct;54(10):2506-14. doi: 10.1007/s00125-011-2204-7. Epub 2011 Jun 9. PMID 21656330
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Unwin N, Rose AMC, George KS, Hambleton IR, Howitt C. The Barbados Health of the Nation Survey: Core Findings. Chronic Disease Research Centre, The University of the West Indies and the Barbados Ministry of Health: St Michael, Barbados, January 2015; 48 pp
- [Background] Karen Bynoe, Maddy Murphy, Charles Taylor, Andre Greenidge, Melissa Abed, Nigel Unwin. The Barbados Diabetes Reversal Study Preliminary Results https://www.cavehill.uwi.edu/fms/resources/cme/78th-cme-presentations/karen-bynoe-barbados-diabetes-reversal-study.aspx
- [Derived] Quimby KR, Murphy MM, Harewood H, Howitt C, Hambleton I, Jeyaseelan SM, Greaves N, Sobers N. Adaptation of a community-based type-2 diabetes mellitus remission intervention during COVID-19: empowering persons living with diabetes to take control. Implement Sci Commun. 2022 Jan 24;3(1):5. doi: 10.1186/s43058-022-00255-9. PMID 35074020
- [Derived] Quimby KR, Sobers N, George C, Greaves N, Browman-Jones F, Samuels TA. Implementation of a community-based low-calorie dietary intervention for the induction of type-2 diabetes and pre-diabetes remission: a feasibility study utilising a type 2 hybrid design. Implement Sci Commun. 2021 Aug 28;2(1):95. doi: 10.1186/s43058-021-00196-9. PMID 34454636